CLINICAL TRIAL: NCT02712073
Title: Predictive Score of the Bowel Preparation Quality Based on a Self-administered Questionnaire
Acronym: PREPA-CO
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Other Study IDs: DRCI V11 01/01/2015
Record Dates: First submitted 2016-03-14; First posted 2016-03-17 (Estimated); Last update posted 2016-04-13 (Estimated); Status verified 2016-04

CONDITIONS: Colonoscopy
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- patients undergoing colonoscopy
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — Self administered questionnaire to evaluate the preparation quality of colonoscopy

SUMMARY:
In France, nearly 1.3 million colonoscopies are performed each year. Colonoscopy is the gold standard in France for colorectal cancer screening in populations at risk. However, it has a number of limitations. The quality of the bowel preparation is a critical step for the successful completion of this examination. The occurrence of interval cancers raises the problem of missed lesions. A literature review showed that there were differences between the endoscopy units on quality standards for bowel preparation. The rate of unprepared colonoscopy is estimated between 20 to 40% . In a recent cohort study, 28% of 2516 colonoscopies had a score of Boston of less than or equal to 6. These colonoscopies generate substantial additional costs to redo colonoscopies, estimated at 35 million euros in 2008. The establishment a predictive score for quality of bowel preparation based on a self-administered questionnaire completed by patients during the pre-colonoscopy consultation, would help identify patients at risk of poor preparation in order to optimize the prescribed preparation in this consultation.

ELIGIBILITY:
Inclusion Criteria:

* Men or woman > 18 years old
* Patient agreeing to participate in the study
* Prescription of a bowel preparation respecting the marketing authorization.

Exclusion Criteria:

* Major patient under guardianship, or protected person,
* Pregnant woman,
* Patient who doesn't understand French or can't read
* People not affiliated with a social security scheme or of such a scheme

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients seen in precolonoscopy consultation
Sampling Method: Non-Probability Sample
Enrollment: 1260 (Estimated)
Dates: Start 2015-05; Primary Completion 2017-09 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
Score performance | within 6 month
  score performance to predict a poor bowel preparation (defined by a score of Boston inferior or equal to 7 and / or a segment equal to 1)

SECONDARY OUTCOMES:
acceptability of questionnaire | end of study
  Acceptability of the questionnaire evaluated by the rate of return of the questionnaires and the rate of well completed questionnaires
Adenoma detection | within 6 month
  adenoma detection rate compared to Boston score

CONTACTS AND LOCATIONS:
Locations (4):
- France (4):
  - Angers UH, Angers
  - Cholet hospital, Cholet
  - La Roche sur Yon hospital, La Roche-sur-Yon
  - Nantes UH, Nantes

IPD SHARING:
Plan to Share IPD: No